CLINICAL TRIAL: NCT05333718
Title: Caracterización de Subgrupos de Diabetes Tipo 2 al diagnóstico: un Paso Necesario Hacia la Medicina de precisión en Diabetes.
Brief Title: Characterization of Type 2 Diabetes Subgroups at Diagnosis: a Necessary Step Towards Precision Medicine in Diabetes.
Acronym: COPERNICAN
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Institut Català de la Salut (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-CDM- 2021-01
Record Dates: First submitted 2022-03-28; First posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Characteristics Disease; Type 2 Diabetes
Keywords: primary care centers; clusters
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Biospecimen Retention: Samples With DNA — blood and urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Newly diagnosed T2DM: To assess and characterize the relevant subgroups (clusters) of type 2 diabetes at diagnosis in our population.
  This objective will be addressed using the 6 main variables that have been used so far in previous studies in other populations to develop disease groupings, that is, age, GAD antibodies, body mass index, glycosylated hemoglobin (HbA1c), and estimates of the evaluation of the homeostatic model 2 of β-cell function and insulin resistance.

SUMMARY:
Objectives: The primary objective is to identify and characterize the relevant subgroups ( clusters ) in type 2 diabetes (T2DM) at the time of diagnosis in our region. This objective will be addressed using the six main variables (see Methodology) used so far in previous studies in other populations to develop the clustering of diabetes. Therefore, this is a study in diagnostic precision medicine in diabetes. In addition, as secondary objectives, other phenotypic characteristics of these subgroups (clinical, metabolic, and associated comorbidities) will be evaluated.

Methodology: This project will establish a prospective observational cohort study of 1200 subjects newly diagnosed with T2DM in primary care centers in the healthcare areas of Barcelona city and the territory of Lleida. All newly diagnosed cases of T2DM will be identified and evaluated. Participants will undergo a comprehensive phenotypic evaluation, including the six variables that will allow the characterization of T2DM subgroups: age, antibodies against glutamic acid decarboxylase (GAD), body mass index, glycated hemoglobin, and sensitivity indices ( HOMA-IR) and insulin secretion (HOMA beta), based on the determination of C-peptide. The latest generation cluster analysis (k- means and hierarchical clustering ) will be performed, following the method described in previous studies using the six variables mentioned above. Onset diabetes subgroups and their association with secondary outcome variables will be assessed. The initial prescription of antidiabetic medication will be evaluated. Other procedures of this project include: clinical (including complications) and biochemical evaluation, advanced lipoprotein profile, and validated questionnaires to evaluate diet and physical activity.

DETAILED DESCRIPTION:
A multicenter prospective observational study will be conducted. The study design contemplates a single visit that will coincide with the inclusion of the patient in the study. Prior to the inclusion visit, a pre-selection period is planned in which the possible candidate will be invited, all the study procedures will be explained and clarified, the selection criteria will be checked and the inclusion visit will be scheduled.

The scope of the study is made up of Primary Care Centers (CAP) in 2 large health areas (Barcelona and Lleida). In the Annex 8 section, the characteristics and expected recruitment capacity of each CAP are detailed. We have taken a conservative approach using the lower range of incidence calculated based on our own data from 2019 to 2020. The table provided used an expected acceptance rate for participation of 80%. Additionally, CAPs were selected based on commitment and performance in our previous studies. It is planned to include 1200 participants newly diagnosed with T2DM. Depending on compliance with the recruitment rate, the inclusion of other CAPs is possible to achieve the expected number of participants in the study.

Follow-up of participants and linkage with other databases

For this study, a pragmatic follow-up of the participants will be chosen, which is adapted to the usual clinical practice for the follow-up of diabetes. For this reason, the monitoring will be done from:

* SIDIAP/PADRIS databases, with the link to the electronic medical record of the participants who have accepted this option in the informed consent.
* Electronic medical record, in the event that the link with the SIDIAP/PADRIS databases is not possible for technical reasons (non-ICS centers), the collection of monitoring variables will be done directly from the clinical course (review of clinical history) of participants without scheduling additional study follow-up visits.
* For specific causes of mortality, data linkage with the National Institute of Statistics (INE) will be used.
* If the participants have already participated or are participating in other clinical research studies and want to transfer the data they have provided for other projects to this study, this linking (portability) of the data will be allowed.

All participants will be followed until the end of the study, death or withdrawal of informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of both sexes, of legal age (≥18 years)
* Newly diagnosed T2DM according to the criteria of the American Diabetes Association
* With a maximum duration of three months of the disease at the time of inclusion.
* Writen informed consent

Exclusion Criteria:

Subjects with a new diagnosis of other types of diabetes (type 1, MODY, gestational or other causes) will also be evaluated to ensure that the diagnostic criteria for selection are correctly implemented in all potential study participants.

*For final analysis, subjects with any diagnosis of diabetes other than T2DM will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with type 2 diabetes mellitus treated in primary care centers in Barcelona and Lleida.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2022-03-08 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
clusters of type 2 diabetes | at inclusion
  To assess and characterize the relevant subgroups (clusters) of type 2 diabetes at diagnosis in our population

SECONDARY OUTCOMES:
gender clinical characteristics | at inclusion
  To assess if there are gender diferences among the type 2 diabetes persons at diagnosis
Frequency of various associated comorbidities, including micro and macrovascular complications | 24 month follow-up period
  To evaluate and describe the complications of type 2 diabetes during the 24 month follow-up period
Advanced lipoprotein profile | at inclusion
  to explore and characterize the lipoprotein profile of the persons with type 2 diabetes at diagnosis
Lifestyle variables: eating habits and physical activity | at inclusion
  to explore if there are differences in lifestyle variables such as eating habits and physical activity at diagnosis of type 2 Diabetes Mellitus
Use in real clinical practice of antidiabetics and other treatments at the beginning of the disease | at inclusion
  to explore if there are differences in treatment of the antidiabetic drugs and other concomitant medications at diagnosis of type 2 Diabetes Mellitus
Appearance of different micro- and macro-vascular complications of diabetes | 24 month follow-up period
  to explore if there are differences in micro and macrovascular complications during the follow-up period related to different sub-types of type 2 Diabetes Mellitus
Metabolomics and genetic profile related to diabetes | at inclusion
  to explore if there are differences in Metabolomics and genetic profile related to different sub-types of type 2 Diabetes Mellitus at diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Dídac Mauricio, MD, PhD, Principal Investigator — Hospital of Santa Creu i Sant Pau
Locations (2):
- Spain (2):
  - Hospital of Santa Creu i Sant Pau, Barcelona, Catalonia
  - Institut Català de la Salut, Barcelona, Catalonia

IPD SHARING:
Plan to Share IPD: No
individual participant data are confidential and will not be shared

REFERENCES:
- [Derived] Fernandez-Camins B, Vlacho B, Canudas A, Ortega M, Granado-Casas M, Perera-LLuna A, Boluda-Sanson A, El-Khattabi-Ofkir Y, Franch-Nadal J, Mauricio D; COPERNICAN Research Group. Characterisation of type 2 diabetes subgroups at diagnosis: the COPERNICAN prospective observational cohort study protocol. BMJ Open. 2024 Dec 15;14(12):e083825. doi: 10.1136/bmjopen-2023-083825. PMID 39675821

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2021-07-17): https://cdn.clinicaltrials.gov/large-docs/18/NCT05333718/Prot_ICF_000.pdf